CLINICAL TRIAL: NCT00920101
Title: Effect of Atorvastatin on Inflammatory Atherosclerotic Plaques Assessed by FDG-PET Imaging
Brief Title: Anti-inflammatory Effect of Atorvastatin in Atherosclerotic Plaques Assessed by FDG-PET Imaging
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Defense Medical College, Japan (Other)
Responsible Party: Principal Investigator, Makoto Ayaori, Assistant Professor, National Defense Medical College, Japan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NDMC570
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Atherosclerosis; Inflammation
Keywords: atherosclerotic plaques; hypercholesterolemia; HMG-CoA reductase inhibitor; statin; lipid-lowering therapy
MeSH Terms: conditions — Atherosclerosis; Inflammation; Plaque, Atherosclerotic; Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Active Comparator)
  Interventions: Drug: Atorvastatin
- Lifestyle counseling (Placebo Comparator): Subjects are advised to keep dietary habits according to the National Cholesterol Education Program (NCEP) from the run-in period throughout the study.
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Drug: Atorvastatin — Subjects are advised to keep dietary habits according to the National Cholesterol Education Program (NCEP) from the run-in period throughout the study. The subjects are administered with 10mg/day for 3 months, if LDL-cholesterol levels does not decrease less than 80mg/dl, the dose is increased up to 20mg/day. If LDL-cholesterol levels decrease less than 60mg/dl, the dose is decreased down to 5mg/day or less.
  Other Names: Lipitor
  Arms: Atorvastatin
Behavioral: Lifestyle counseling — Subjects are advised to keep dietary habits according to the National Cholesterol Education Program (NCEP) from the run-in period throughout the study.
  Arms: Lifestyle counseling

SUMMARY:
The purpose of this study is to determine whether HMG-CoA reductase inhibitor, atorvastatin attenuates inflammation in atherosclerotic plaques detected by 18F-fluorodeoxyglucose(FDG) PET.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with accumulation of FDG-PET in carotid artery or aorta

Exclusion Criteria:

* LDL cholesterol level (calculated by using Friedewald formula) higher than 180 mg/dl or less than 120 mg/dl
* subjects currently taking HMG CoA-reductase (Statins) or fibrates
* symptomatic coronary artery diseases
* symptomatic cerebrovascular diseases
* subjects suffered from myocardial infarction or stroke within 6 months
* subjects underwent percutaneous vascular interventions or vascular operations within 6 months
* diabetic patients with poor glycemic control (HbA1c>8.5)
* hypertensive patients with poor blood pressure control
* subjects with neoplasms
* subjects with systemic inflammatory diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) of 18-FDG detected in carotid/aortic atherosclerotic plaques | Baseline and 3 months after intervention

SECONDARY OUTCOMES:
Flow-mediated vasodilation of brachial artery determined by ultrasonography | Baseline and 3 months after intervention
Serum markers for inflammation such as high-sensitive CRP, IL-6 or soluble ICAM-1 | Baseline and 3 months after intervention
Serum and urine markers for anti- or pro-oxidant stress such as oxidized LDL or 8-Hydroxydeoxyguanosine | Baseline and 3 months after intervention
Max-intima-media thickness (Max-IMT), Mean-IMT and plaque score determined by carotid artery ultrasonography | Baseline and 3 months after intervention
Serum lipids such as total cholesterol, LDL-cholesterol, HDL-cholesterol, RLP-cholesterol and triglycerides | Baseline and 3 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Katsunori Ikewaki, Principal Investigator — National Defense Medical College
Locations (1):
- National Defense medical College, Tokotozawa, Saitama, Japan